CLINICAL TRIAL: NCT03324906
Title: Effects of Transcranial Direct Current Stimulation (tDCS) on Obsessive Compulsive Behavior and Depressive Symptoms on Individuals With Prader-Willi Syndrome
Brief Title: Effects of Transcranial Direct Current Stimulation (tDCS) on Individuals With Prader-Willi Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Caroline Azevedo, Especialist, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 58280016.1.0000.5505
Record Dates: First submitted 2017-10-08; First posted 2017-10-30 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Prader-Willi Syndrome; Obesity; Depressive Disorder; Obsessive-Compulsive Disorder
Keywords: Prader-Willi Syndrome; Obesity; Depressive disorder; Obsessive-compulsive disorder; noninvasive brain stimulation
MeSH Terms: conditions — Prader-Willi Syndrome; Obesity; Depressive Disorder; Obsessive-Compulsive Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tDCS active Prader-Willi Syndrome (Active Comparator): The anode will be placed in the left side of DLPFC (F3) of the International Electrode Placement System 10-20 and cathode will be placed in the same region of the contralateral cortex, corresponding to the area F4. The stimulation current will be 2mA (for individuals aged 14-35 years) and 1mA (for individuals aged 11 to 13 years, maintaining this intensity until the end of the stimulation), will last for thirty seconds, and the ramp will exit fifteen seconds. The stimulation will last for up to 20 minutes, for a total of 10 sessions, one a day for twice a week with a weekend break.
  Interventions: Device: tDCS
- tDCS active Obese Subjects (Active Comparator): The stimulation current will be 2mA (for individuals aged 14-35 years) and 1mA (for individuals aged 11 to 13 years, maintaining this intensity until the end of the stimulation). The start ramp, when the current will be changed from zero to 2mA (two milli amps), will last for thirty seconds, and the ramp will exit fifteen seconds. The stimulation will last for up to 20 minutes.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — The anode will be placed in the left side of DLPFC (F3) of the International Electrode Placement System 10-20 and cathode will be placed in the same region of the contralateral cortex, corresponding to the area F4. The stimulation current will be 2mA (for individuals aged 14-35 years) and 1mA (for individuals aged 11 to 13 years, maintaining this intensity until the end of the stimulation), will last for thirty seconds, and the ramp will exit fifteen seconds. The stimulation will last for up to 20 minutes, for a total of 10 sessions, one a day for twice a week with a weekend break.
  Other Names: There aren't others interventions

SUMMARY:
Prader-Willi Syndrome (PWS) is a multisystemic genetic disease characterized by hypotonia, mental retardation, hyperphagia, and uncontrollable hunger due to hypothalamic dysfunction, caused by dysregulation of genes located in chromosome 15q11-q13. The goal of this study is to evaluate the effects of Transcranial Direct Current Stimulation (tDCS) on hyperphagia and behavior in PWS. Forty children and adolescents (11-24 years) with clinical and cytogenetic-molecular diagnosis of Prader-Willi syndrome will be assessed before and after 10 tDCS session with: Food Craving Questionnaire (FCQ), Aberrant Behavior Checklist (ABC), Dykens hyperphagia questionnaire. Caregivers self-reported the participant's behaviors at home and, lately, they will be categorized and quantified. tDCS will be applied for 20 minutes with electrodes of 25cm2 wrapped in cotton material soaked in saline solution. The anode at the left dorsolateral prefrontal cortex (F3) and the cathode at the contralateral area (F4). Children from 11-12 years will receive a current of 1mA; above 13 years, 2mA.

DETAILED DESCRIPTION:
Prader-Willi syndrome (PWS) is a complex neurodevelopmental disorder that affects about 1 in 20,000 births, regardless of sex or race. PWS is characterized by two clinical phases. In the first, the cardinal symptoms are: neonatal hypotonia, feeding difficulty, lethargy, weak crying and hyporeflexia. The second, from six months, presents gradual improvement of hypotonia, weight gain and progressive development of hyperphagia and obesity. A recent trend is the use of transcranial Direct Current Stimulation (tDCS), a very simple, safe and inexpensive technique of cerebral stimulation, noninvasive and painless. It is based on the application of low intensity direct current (0-2 mA) through electrodes. tDCS has been shown to be a safe, easily tolerable method, allowing its therapeutic use in several clinical situations involving sustained cortical dysfunction such as in neurological or psychiatric disorders, including Schizophrenia, Alzheimer's Disease, Parkinson's Disease and major depression. These and other studies have been shown to be consistent with tDC's therapeutic methodology, thus favoring more accurate conclusions about the efficacy and efficiency of the method. The general objective of this research is to evaluate the effects of tDCS on the treatment Obsessive Compulsive Behavior and depressive symptoms in PWS; evaluate and compare the participants' cerebral activation pattern through electroencephalographic mapping with resting-quantitative EEG (qEEG), before and after the intervention; check if the changes (if any) last 3 months after the end of the intervention (follow up). 40 individuals will be invited to participate in this study, divided into 2 groups: 20 patients with PWS, in the age group between 11 and 35 years of age diagnosed and 20 obese individuals without the diagnosis of PWS. All will receive the same pacing protocol in terms of number of sessions and pacing time, tDCS intensity will be adjusted to 1mA in subjects aged 11 to 13 years and up to 2mA in subjects aged 14-35 years. The project will include Neuropsychological evaluation for each patient and electroencephalographic mapping with resting qEEG, before and after the intervention at the beginning of the experiment, at the end of the experiment and 30 days after (follow up).

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged above 11 years old;
* BMI > 30Kg/m²
* Agreement and Consent of parents and/or guardians and adolescent to participate of the study.

Exclusion Criteria:

* Cognitive inability to understand instructions, as assessed by the psychiatrist, due to severe cognitive impairment;
* Presence of other associated syndromes in addition to PWS;
* Inability to travel to the research site due to complications due to obesity; for convenience, as they seek specialized centers for the care of this population and associations of Prader Willi they will be referred by those responsible for participation in the program.

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-05-08 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Hyperphagia changes | This outcome will be evaluate at the baseline [T1], 10 days after baseline - last stimulation session [T2] and 30 days of follow up [T3].
  We expect changes in hyperphagic behaviors assessed by the Dykens Scale. This is a 13-item instrument that was specifically designed to measure food-related pre-occupations and problems in PWS, as well as the severity of these concerns. Items reflected parent and offspring reports of hyperphagic symptoms gleaned from our ongoing research and clinic programs for persons with PWS and their families. The severity items were based on the definition of symptom-related impairment as operationalized by the American Psychiatric Association. Items on the Dikens Scale were rated on a five-point scale (1 = not a problem to 5 = severe and/or frequent problem). The final score will be defined as the sum of all subscales. The higher is this score, the worse is the outcome.

SECONDARY OUTCOMES:
Improve depressive symptoms | This outcome will be evaluate at the baseline [T1], 10 days after baseline - last stimulation session [T2] and 30 days of follow up [T3].
  We expect to improve depressive symptoms assessed by the Beck Depression Inventory (BDI). This is a 21-item self-report inventory, which assess depressive symptoms in the last seven days. The cut-off point for this scale is defined by: <10 = no symptoms of depression; 10 - 18 = slight to moderate symptoms of depression; 19 - 29 = moderate to severe symptoms of depression; and 30 - 63 = severe symptoms of depression. The final score will be defined based on the sum of all subscales. The higher is this score, the worse is the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Azevedo, especialist, Principal Investigator — Federal University of São Paulo
Locations (1):
- Caroline Azevedo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Azevedo C, Gomes JS, Trevizol AP, Dias AM, Cordeiro Q. At-Home Transcranial Direct Current Stimulation in Prader-Willi Syndrome With Severe Intellectual Disability: A Case Study. J ECT. 2017 Sep;33(3):e29-e30. doi: 10.1097/YCT.0000000000000409. No abstract available. PMID 28383347